CLINICAL TRIAL: NCT01663727
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study To Evaluate the Efficacy and Safety Of Bevacizumab, and Associated Biomarkers, In Combination With Paclitaxel Compared With Paclitaxel Plus Placebo as First-line Treatment Of Patients With Her2-Negative Metastatic Breast Cancer
Brief Title: Study To Evaluate the Efficacy and Safety Of Bevacizumab, and Associated Biomarkers, In Combination With Paclitaxel Compared With Paclitaxel Plus Placebo as First-line Treatment Of Patients With Her2-Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GO25632; 2011-005335-97 (EudraCT Number)
Record Dates: First submitted 2012-08-09; First posted 2012-08-13 (Estimated); Results first posted 2016-02-10 (Estimated); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental): Paclitaxel + Bevacizumab [Avastin]
  Interventions: Drug: Bevacizumab [Avastin]; Drug: Paclitaxel
- B (Experimental): Paclitaxel + Placebo
  Interventions: Drug: Paclitaxel; Drug: Placebo

INTERVENTIONS:
Drug: Bevacizumab [Avastin] — Intravenous repeating dose
  Arms: A
Drug: Paclitaxel — Intravenous repeating dose
Drug: Placebo — Intravenous repeating dose
  Arms: B

SUMMARY:
This is a Phase III, randomized, double-blind, placebo-controlled multicenter study to evaluate the efficacy and safety of bevacizumab administered in combination with paclitaxel in patients with previously untreated, locally recurrent, or metastatic HER2-negative breast cancer. Patients will be randomized to one of two treatment arms: bevacizumab or placebo. All patients will be given an intravenous (IV) infusion of of paclitaxel (90 mg/m2) for 3 weeks during each 28-day cycle. bevacizumab or placebo (10 mg/kg) will be administered by IV infusion on Days 1 and 15 of each 28-day cycle. Patients will be treated until disease progression, unacceptable toxicity or death from any cause occurs.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed, HER2-negative adenocarcinoma of the breast, with measurable or non-measurable locally recurrent or metastatic disease. Locally recurrent disease must not be amenable to resection with curative intent.
* ECOG performance status of 0 or 1
* For women of childbearing potential, use of an acceptable and effective method of non-hormonal contraception
* For patients who have received recent radiotherapy, recovery prior to randomization from any significant acute toxicity, and radiation treatments have to be completed more than 3 weeks from randomization

Exclusion Criteria:

Disease-Specific Exclusions:

* HER2-positive status
* Prior chemotherapy for locally recurrent or metastatic disease
* Prior hormonal therapy < 2 weeks prior to randomization
* Prior adjuvant or neo-adjuvant chemotherapy is allowed, provided its conclusion has been for at least 12 months prior to randomization
* Investigational therapy within 28 days of randomization

General Medical Exclusions:

* Life expectancy of < 12 weeks
* Inadequate organ function
* Uncontrolled serious medical or psychiatric illness
* Active infection requiring intravenous (IV) antibiotics at screening
* Pregnancy or lactation
* History of other malignancies within 5 years prior to screening, except for tumors with a negligible risk for metastasis or death

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 481 (Actual)
Dates: Start 2012-08-27 (Actual); Primary Completion 2014-11-30 (Actual); Study Completion 2017-11-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (177):
- United States (65):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - Wilshire Oncology Medical Group, Corona, California
  - Wilshire Oncology Medical Group, Glendora, California
  - Wilshire Oncology Medical Group, La Verne, California
  - Long Beach Memorial Medical Center; Oncology, Long Beach, California
  - Tenet Health System Desert Inc, Palm Springs, California
  - Wilshire Oncology Medical Group; Oncology, Pomona, California
  - Wilshire Oncology Medical Group, Rancho Cucamonga, California
  - Wilshire Oncology Medical Group, West Covina, California
  - Washington Hospital, Washington D.C., District of Columbia
  - Sylvester Comprehensive Cancer Center - Deerfield Beach; Sylvester Cancer Center, Deerfield Beach, Florida
  - Florida Cancer Specialists - Broadway, Fort Myers, Florida
  - BRCR Medical Center, Inc., Plantation, Florida
  - Hematology Oncology Associates of the Treasure Coast, Port Saint Lucie, Florida
  - Northeast Georgia Cancer Care LLC, Athens, Georgia
  - Peachtree Hematology & Oncology Consultants, Pc, Atlanta, Georgia
  - Kaiser Foundation Hospital; Dr. Eron's Office, Honolulu, Hawaii
  - IU Cancer Pavilion, Indianapolis, Indiana
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Lahey Clinic Inc. - PARENT ACCOUNT, Burlington, Massachusetts
  - The Jones Clinic, PC, New Albany, Mississippi
  - Missouri Cancer Associates, Columbia, Missouri
  - Washington University; Center for Adv Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Signal Point Clinical; Research Center, LLC, Middletown, Ohio
  - ProMedica Hickman Cancer Center at Flower Hospital; Hickman Cancer Center, Sylvania, Ohio
  - University of Toledo; Dept. of Medicine, Toledo, Ohio
  - Virginia Cancer Specialists - Leesburg, Leesburg, Pennsylvania
  - Pennsylvania Oncology Hematology Associates, Inc.; PA Oncology & Hematology, Philadelphia, Pennsylvania
  - Medical University of South Carolina; Division of Hematology-Oncology, Charleston, South Carolina
  - SCRI-Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology-Medical City Dallas, Dallas, Texas
  - Texas Oncology, P.A. - Dallas Presbyterian, Dallas, Texas
  - Texas Oncology, P.A. - Fort Worth, Fort Worth, Texas
  - Texas Oncology- Southwest Fort Worth, Fort Worth, Texas
  - Univ of Texas Medical Branch, Galveston, Texas
  - Texas Oncology, P.A. - Garland, Garland, Texas
  - Cancer Care Centers of S Texas, Kerrville, Texas
  - Texas Oncology- Longview Cancer Center, Longview, Texas
  - Texas Oncology, P.A. - McAllen; South Texas Cancer Center-McAllen, McAllen, Texas
  - Texas Oncology Plano West, Plano, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - CancerCare Centers of South Texas, San Antonio, Texas
  - Texas Oncology, P.A. - Tyler, The Woodlands, Texas
  - Texas Oncology, P.A., The Woodlands, Texas
  - Virginia Cancer Specialists - Alexandria, Alexandria, Virginia
  - Fairfax Northern Virginia Hematology-Oncology PC, Arlington, Virginia
  - Wellmonth Physician Services, Bristol, Virginia
  - Virginia Oncology Associates - Chesapeake, Chesapeake, Virginia
  - Oncology & Hematology Associates of SW Va Inc. - Market Street, Christiansburg, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Hematology Oncology Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Virginia Cancer Specialists - Gainsville, Gainesville, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Oncology and Hematology Assoc. of SW VA, Inc. - Low Moor, Low Moor, Virginia
  - Virginia Oncology Associates - New Port News, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Oncology & Hematolgy Associates of SW Va Inc. - Roanoke, Roanoke, Virginia
  - Oncology and Hematology Assoc. of SW VA, Inc., Salem, Virginia
  - Virginia Oncology Associates - Virginia Beach, Virginia Beach, Virginia
  - Oncology and Hematology Assoc. of SW VA, Inc. - Wytheville, Wytheville, Virginia
  - Northwest Medical Specialties, PLLC; Research Department, Tacoma, Washington
  - West Virginia University; Endocrinology, Morgantown, West Virginia
- Argentina (9):
  - Hospital Britanico de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Centro de Investigacion Pergamino SA, Pergamino
  - Instituto de Investigaciones Clínicas Quilmes, Quilmes
  - Hospital Provincial del Centenario, Rosario
  - Instituto CAICI, Rosario
  - Instituto de Oncología de Rosario, Rosario
  - Sanatorio Parque S.A., Rosario, Santa FE
  - ISIS Clinica Especializada, Santa Fe
- Belgium (5):
  - AZ KLINA, Brasschaat
  - UZ Brussel, Brussels
  - UZ Antwerpen, Edegem
  - GHdC Site Saint-Joseph, Gilly (Charleroi)
  - CHU Ambroise Paré; Hematology and Oncology Department, Mons
- Brazil (9):
  - Clinica de Tratamento e Pesquisa Oncologica - Oncotek, Brasília, Federal District
  - Hospital da Cidade de Passo Fundo; Centro de Pesquisa em Oncologia, Passo Fundo, Rio Grande do Sul
  - Hospital Sao Lucas - PUCRS; Pesquisa Clinica, Porto Alegre, Rio Grande do Sul
  - Clinica de Oncologia de Porto Alegre - CliniOnco, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Hospital das Clinicas - FMUSP Ribeirao Preto, Ribeirão Preto, São Paulo
  - Universidade Federal de Sao Paulo - UNIFESP, São Paulo, São Paulo
- Bulgaria (10):
  - MHAT Dr. Tota Venkova AD, Gabrovo
  - SHATOD Haskovo EOOD, Haskovo
  - Complex Oncological Center - Plovdiv, EOOD, Plovdiv
  - Complex Oncological Center - Shumen, EOOD; Department of Chemotherapy, Shumen
  - SHATOD - Sofia District, EOOD, Sofia
  - MHAT Serdika, EOOD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL, EAD, Sofia
  - SHATOD - Sofia City, EOOD, Sofia
  - SHATOD Dr. Marko Antonov Markov-Varna, EOOD, Varna
  - COC - Veliko Tarnovo, Veliko Tarnovo
- Chile (4):
  - Centro de Estudios Oncologicos de Santiago (CEOS) Oncologia, Santiago
  - Fundacion Arturo Lopez Perez, Santiago
  - Instituto Nacional del Cancer, Santiago
  - Instituto Oncologico Ltda., Viña del Mar
- Germany (6):
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - St. Elisabeth-Krankenhaus, Cologne
  - St. Johannes Hospital; Klinik fuer innere Medizin II, Onkologie, Haematologie, Dortmund
  - Wilhelm-Anton-Hospital gGmbH, Goch
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitaetsklinikum Ulm, Ulm
- Italy (7):
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera A. Cardarelli, Napoli, Campania
  - Ospedale degli Infermi, Rimini, Emilia-Romagna
  - Ospedale Mater Salutis, Legnago (VR), Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Fondazione Salvatore Maugeri IRCCS, Pavia, Lombardy
  - Ospedale Versilia, Lido di Camaiore, Tuscany
- Japan (20):
  - NHO Shikoku Cancer Center; Dept of Respiratory Medicine, Ehime
  - NHO Kyushu Cancer Center, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima University Hospital, Hiroshima
  - Hyogo College of Medicine Hospital, Hyōgo
  - Hakuaikai Sagara Hospital, Kagoshima
  - Tokai University Hospital, Kanagawa
  - Kumamoto University Hospital, Kumamoto
  - Kumamoto City Hospital, Kumamoto
  - Tohoku University Hospital, Miyagi
  - Niigata Cancer Center Hospital, Niigata
  - Iwate Medical University Hospital, Numakunai
  - NHO Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Osaka
  - NHO Hokkaido Cancer Center, Sapporo
  - Shizuoka General Hospital, Shizuoka
  - Toranomon Hospital, Tokyo
  - Juntendo University Hospital, Tokyo
  - Tokyo Metropolitan Cancer and Infectious diseases Center Komagome Hospital, Tokyo
- Panama (2):
  - Centro Hemato Oncologico Panama, Panama City
  - Medical Research Centre, Panama City
- Romania (4):
  - Institutul Oncologic "Prof. Dr. Al. Trestioreanu", Bucharest
  - Institutul Oncologic Prof. Dr. Ion Chiricuta Cluj-Napoca; Radioterapie I - Oncologie, Cluj-Napoca
  - Medisprof SRL, Cluj-Napoca
  - Oncomed SRL, Timișoara
- Russia (9):
  - CTPI Chernihiv Regional Oncological Dispensary, Chernihiv
  - SHI Republican Clinical Oncological Dispensary of HM RT, Kazan'
  - Regional Clinical Oncology Dispensary, Krasnodar
  - FSBSI "Russian Oncological Scientific Center n.a. N.N. Blokhin", Moscow
  - Non-state Healthcare Institution "Road Clinical Hospital of JSC Russian Railways", Saint Petersburg
  - City Clinical Oncology Dispensary, Saint Petersburg
  - SBEIHPE SSMU n.a. I.P.Pavlov of MOH and SD of RF, Saint Petersburg
  - FBI "Scientific Research Institute of Oncology n. a. N. N. Petrov", Saint Petersburg
  - Samara Regional Oncology Dispensary, Samara
- South Africa (7):
  - National Hospital; Oncotherapy Dept, Bloemfontein
  - Cape Town Oncology Trials, Cape Town
  - Hopelands Cancer Centre Durban, Durban
  - Mary Potter Oncology Centre, Groenkloof
  - Hopelands Cancer Centre, Hilton
  - Cancercare, Port Elizabeth
  - University of Pretoria; Department of Medical Oncology, Pretoria
- South Korea (6):
  - National Cancer Centre, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System; Pharmacy, Seoul
  - Asan Medical Center., Seoul
  - Samsung Medical Center, Seoul
- Ukraine (8):
  - CI Cherkasy Regional Oncological Dispensary of Cherkasy RC RC of Clinical Oncology, Cherkassy
  - CI Dnipropetrovsk CMCH 4 of Dnipropetrovsk RC Dept of Chemotherapy SI Dnipropetrovsk MA of MOHU, Dnipropetrovsk
  - CCTPI Donetsk Regional Antitumor Center, Donetsk
  - Kyiv Сity Clinical Oncological Center, Kyiv
  - Medical and Prophylactic Institution Volyn Regional Oncological Dispensary, Lutsk
  - Lviv State Oncological Regional Treatment and Diagnostic Center, Lviv
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
  - CCCH City Oncological Center SHEI Uzhgorod NU, Uzhhorod
- United Kingdom (6):
  - Velindre Cancer Centre, Cardiff
  - Western General Hospital, Edinburgh
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Mount Vernon Hospital, Middlesex
  - Peterborough City Hospital, Peterborough
  - Derriford Hospital; Clinical Neurology Research Group, Plymouth

REFERENCES:
- [Derived] Masuda N, Takahashi M, Nakagami K, Okumura Y, Nakayama T, Sato N, Kanatani K, Tajima K, Kashiwaba M. First-line bevacizumab plus paclitaxel in Japanese patients with HER2-negative metastatic breast cancer: subgroup results from the randomized Phase III MERiDiAN trial. Jpn J Clin Oncol. 2017 May 1;47(5):385-392. doi: 10.1093/jjco/hyx001. PMID 28158579
- [Derived] Miles D, Cameron D, Bondarenko I, Manzyuk L, Alcedo JC, Lopez RI, Im SA, Canon JL, Shparyk Y, Yardley DA, Masuda N, Ro J, Denduluri N, Hubeaux S, Quah C, Bais C, O'Shaughnessy J. Bevacizumab plus paclitaxel versus placebo plus paclitaxel as first-line therapy for HER2-negative metastatic breast cancer (MERiDiAN): A double-blind placebo-controlled randomised phase III trial with prospective biomarker evaluation. Eur J Cancer. 2017 Jan;70:146-155. doi: 10.1016/j.ejca.2016.09.024. Epub 2016 Nov 4. PMID 27817944

RESULTS

PARTICIPANT FLOW:
Groups:
- Paclitaxel+Placebo: Participants received paclitaxel 90 mg/m^2 IV on Days 1, 8 and 15 and placebo matched to bevacizumab IV infusion on Days 1 and 15 of a 28 day cycle until progressive disease, treatment limiting toxicity or death.
- Paclitaxel+ Bevacizumab: Participants received paclitaxel 90 mg/m^2 IV on Days 1, 8 and 15 and bevacizumab IV 10 mg/kg on Days 1 and 15 of a 28 day cycle until progressive disease, treatment limiting toxicity or death.
Period: Overall Study
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Started | 242 | 239
Completed | 0 | 1
Not Completed | 242 | 238
Not completed — Death | 161 | 155
Not completed — Lost to Follow-up | 10 | 8
Not completed — Withdrawal by Subject | 18 | 25
Not completed — Study Terminated | 51 | 50
Not completed — Withdrawal by subject and Adverse Event. | 1 | 0
Not completed — Withdrawal prior to dosing. | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All participants randomized to study treatment irrespective of whether the assigned treatment was actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab | Total
Number analyzed (Participants) | 242 | 239 | 481
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (10.7) | 55.8 (11.5) | 55.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 237 | 236 | 473
  Male | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression or Death in Intent-to-Treat (ITT) Population
Description: Tumor assessment was performed as per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) by investigator. Disease progression was defined as at least 20 percent (%) increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 millimeter (mm), unequivocal progression of existing non-target lesions, or presence of new lesions.
Time Frame: Baseline, every 8 weeks until documented disease progression, death or clinical cut-off (up to 117.7 weeks)
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 242 | 239
percentage of participants | 69.4 | 63.6

2. Primary Outcome: Progression Free Survival (PFS) in ITT Population
Description: PFS was defined as the interval between the date of randomization and the first documentation of progressive disease or death from any cause. Tumor assessment was performed as per RECIST v1.1 by investigator. Disease progression was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, unequivocal progression of existing non-target lesions, or presence of new lesions. PFS was estimated using Kaplan Meier method.
Time Frame: Baseline, every 8 weeks until documented disease progression, death or clinical cut-off (up to 117.7 weeks)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 242 | 239
months | 8.8 [7.4 to 9.3] | 11.0 [9.5 to 12.2]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Stratified analysis: Stratification factors were plasma VEGF-A level (low/high), prior adjuvant chemotherapy (yes/no) and estrogen receptor / progesterone receptor status (positive, negative); Test type: Superiority or Other; p = 0.0007, Log Rank; Hazard Ratio (HR) = 0.68, 99% CI 2-sided [0.51 to 0.91] — Hazards ratio was estimated by Cox regression
Statistical Analysis 2: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Unstratified Analysis; Test type: Superiority or Other; p = 0.0046, Log Rank; Hazard Ratio (HR) = 0.73, 99% CI 2-sided [0.55 to 0.97]
Statistical Analysis 3: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; A stratified multivariate Cox regression model, including treatment, VEGF-A level, and interaction between treatment and VEGF-A level (low, high) as factors was used to estimate the interaction p-value of the treatment with VEGF-A level for PFS. Analysis for the interaction of treatment effect with the plasma VEGF-A levels was a secondary objective; Test type: Superiority or Other; p = 0.4619, Wald Test

3. Secondary Outcome: Percentage of Participants Who Died - ITT Population
Time Frame: From randomization till death or clinical cut-off (up to 244 weeks)
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 242 | 239
percentage of participants | 64.9 | 64.0

4. Secondary Outcome: Overall Survival (OS) - ITT Population
Description: OS was defined as the interval between the date of randomization and death from any cause. OS was estimated using Kaplan Meier method.
Time Frame: From randomization till death or clinical cut-off (up to 244 weeks)
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 242 | 239
months | 25.8 [21.8 to 30.2] | 28.8 [22.8 to 32.8]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Stratified analysis: Stratified analysis: Stratification factors were plasma VEGF-A level (low/high), prior adjuvant chemotherapy (yes/no) and estrogen receptor / progesterone receptor status (positive, negative); Test type: Superiority or Other; p = 0.5877, Log Rank; Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.75 to 1.18] — Hazards ratio was estimated by Cox regression
Statistical Analysis 2: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Unstratified analysis; Test type: Superiority or Other; p = 0.8004, Log Rank; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.78 to 1.21] — Hazards ratio was estimated by Cox regression

5. Secondary Outcome: Percentage of Participants Who Died - High Baseline Plasma VEGF-A ITT Population
Time Frame: From randomization till death or clinical cut-off (up to 244 weeks)
Population: High Baseline Plasma VEGF-A ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 124 | 120
percentage of participants | 74.2 | 71.1

6. Secondary Outcome: OS - High Baseline Plasma VEGF-A ITT Population
Description: as for outcome 4
Time Frame: From randomization till death or clinical cut-off (up to 244 weeks)
Population: High Baseline Plasma VEGF-A ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 124 | 120
months | 19.4 [16.5 to 25.0] | 22.8 [18.2 to 31.6]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Stratified analysis: Stratification factors were prior adjuvant chemotherapy (yes/no) and estrogen receptor / progesterone receptor status (positive, negative); Test type: Superiority or Other; p = 0.2745, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.63 to 1.14] — Hazards ratio was estimated by Cox regression
Statistical Analysis 2: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Unstratified analysis; Test type: Superiority or Other; p = 0.3616, Log Rank; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.65 to 1.17] — Hazards ratio was estimated by Cox regression

7. Secondary Outcome: Percentage of Participants With an Objective Response - ITT Population
Description: Objective response was defined as having a Complete Response (CR) or Partial Response (PR) according to a RECIST criteria v 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Measurable disease was defined by the presence of at least one measurable lesion by clinical measurement, chest x-ray, computed tomography (CT), or magnetic resonance imaging (MRI).
Time Frame: Baseline, every 8 weeks until documented disease progression, death or clinical cut-off (up to 117.7 weeks)
Population: Number of participants analyzed=participants from ITT population with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 214 | 202
percentage of participants | 33.2 [26.87 to 39.49] | 54.0 [47.09 to 60.83]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Test type: Superiority or Other; p < 0.0001, Fisher; Difference in Response Rates = 20.78, 95% CI 2-sided [11.45 to 30.11]

8. Primary Outcome: Percentage of Participants With Progression or Death in High Baseline Plasma Vascular Endothelial Growth Factor-A (VEGF-A) ITT Population
Description: Tumor assessment was performed as per RECIST v1.1 by investigator. Disease progression was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, unequivocal progression of existing non-target lesions, or presence of new lesions.
Time Frame: Baseline, every 8 weeks until documented disease progression, death or clinical cut-off (up to 111.3 weeks)
Population: High baseline plasma VEGF-A ITT population: All participants randomized to study treatment with high baseline plasma VEGF-A levels (VEGF-A levels greater than or equal to 5.05 picograms per milliliter), irrespective of whether the assigned treatment was actually received.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 124 | 120
percentage of participants | 75.0 | 70.8

9. Primary Outcome: PFS in High Baseline Plasma VEGF-A ITT Population
Description: as for outcome 2
Time Frame: Baseline, every 8 weeks until documented disease progression, death or clinical cut-off (up to 111.3 weeks)
Population: High baseline plasma VEGF-A ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 124 | 120
months | 7.3 [5.6 to 8.7] | 9.6 [9.0 to 11.0]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.0038, Log Rank; Hazard Ratio (HR) = 0.64, 96% CI 2-sided [0.47 to 0.88] — Hazards ratio was estimated by Cox regression
Statistical Analysis 2: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Unstratified analysis; Test type: Superiority or Other; p = 0.0101, Log Rank; Hazard Ratio (HR) = 0.68, 96% CI 2-sided [0.50 to 0.93]

10. Secondary Outcome: Percentage of Participants With an Objective Response - High Baseline Plasma VEGF-A ITT Population
Description: Objective response was defined as having a CR or PR according to a RECIST criteria v 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Measurable disease was defined by the presence of at least one measurable lesion by clinical measurement, chest x-ray, CT, or MRI.
Time Frame: Baseline, every 8 weeks until documented disease progression, death or clinical cut-off (up to 111.3 weeks)
Population: Number of participants analyzed=participants from high baseline plasma VEGF-A ITT population with measurable disease at baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 116 | 105
percentage of participants | 32.8 [24.22 to 41.30] | 54.3 [44.76 to 63.81]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Test type: Superiority or Other; p = 0.0017, Fisher; Difference in Response Rates = 21.53, 95% CI 2-sided [8.73 to 34.32]

11. Secondary Outcome: Duration of Response - ITT Population
Description: Duration of response was defined as the time from the initial date of the objective response to documented disease progression or death (whichever occurred first). Objective response was defined as having a CR or PR according to a RECIST criteria v 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Disease progression was defined as at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, unequivocal progression of existing non-target lesions, or presence of new lesions. Analysis was performed using Kaplan Meier method.
Time Frame: Baseline, every 8 weeks until documented disease progression or clinical cut-off (up to 117.7 weeks)
Population: Number of participants analyzed=participants from ITT population who had an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 71 | 109
months | 9.2 [7.4 to 11.5] | 9.5 [7.8 to 12.4]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.2737, Log Rank; Hazard Ratio (HR) = 0.80, 95% CI 2-sided [0.54 to 1.19] — Hazards ratio was estimated by Cox regression
Statistical Analysis 2: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Unstratified analysis; Test type: Superiority or Other; p = 0.2959, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.56 to 1.19] — Hazards ratio was estimated by Cox regression

12. Secondary Outcome: Duration of Response - High Baseline Plasma VEGF-A ITT Population
Description: Duration of response was defined as the time from the initial date of the objective response to documented disease progression or death (whichever occurred first). Objective response was defined as having a CR or PR according to a RECIST criteria v 1.1. CR was defined as disappearance of all target and non-target lesions and no new lesions, all pathological lymph nodes must have decreased to <10 mm in short axis and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions (taking as reference the baseline sum diameters), no progression in non-target lesions, and no new lesions. Disease progression was defined at least 20% increase in the sum of diameters of target lesions compared to smallest sum of diameters on-study and absolute increase of at least 5 mm, unequivocal progression of existing non-target lesions, or presence of new lesions. Analysis was performed using Kaplan Meier method.
Time Frame: Baseline, every 8 weeks until documented disease progression or clinical cut-off (up to 111.3 weeks)
Population: Number of participants analyzed=participants from high baseline plasma VEGF-A ITT population who had an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 38 | 57
months | 7.2 [5.6 to 9.5] | 8.1 [7.1 to 11.1]
Statistical Analysis 1: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.1783, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.41 to 1.18] — Hazards ratio was estimated by Cox regression
Statistical Analysis 2: Comparison: Paclitaxel+Placebo vs Paclitaxel+ Bevacizumab; Unstratified analysis; Test type: Superiority or Other; p = 0.2429, Log Rank; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.45 to 1.22] — Hazards ratio was estimated by Cox regression

13. Secondary Outcome: Percentage of Participants Who Were Alive at 1 Year - ITT Population
Time Frame: 1 year
Population: ITT Population.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 242 | 239
percentage of participants | 80.94 | 82.47

14. Secondary Outcome: Secondary: Percentage of Participants Who Were Alive at 1 Year - High Baseline Plasma VEGF-A ITT Population
Time Frame: 1 year
Population: High Baseline Plasma VEGF-A ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
Number analyzed (Participants) | 124 | 120
percentage of participants | 69.27 | 80.96

ADVERSE EVENTS:
Time Frame: From the first dose of study drug through 30 days after the last dose of study drug or clinical cut-off (up to 115.1 weeks)
Description: Safety population: All randomized participants who received at least one full or partial dose of any component of the study treatment (bevacizumab, placebo, or paclitaxel).
Arm/Group | Paclitaxel+Placebo | Paclitaxel+ Bevacizumab
All-Cause Mortality (participants affected / at risk) | 162/233 | 161/238
Serious Adverse Events (participants affected / at risk) | 45/233 | 66/238
Other Adverse Events (participants affected / at risk) | 225/233 | 230/238
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel+Placebo (N=233) | Paclitaxel+ Bevacizumab (N=238)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 1 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Optic nerve disorder (Eye disorders) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (6) | 2 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 4 (4)
Asthenia (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 1 (3) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 3 (3)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 4 (6)
Cholecystitis infective (Infections and infestations) | 0 (0) | 1 (1)
Colonic abscess (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 2 (2) | 3 (3)
Device related sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (4) | 4 (4)
Pneumonia necrotising (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis syndrome (Infections and infestations) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2)
Wound infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Urine output decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 3 (4)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Embolism venous (Vascular disorders) | 1 (1) | 0 (0)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 1 (1)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
CATARACT (Eye disorders) | 1 (1) | 0 (0)
CATHETER SITE ERYTHEMA (General disorders) | 0 (0) | 1 (2)
ANAPHYLACTIC REACTION (Immune system disorders) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
CATHETER SITE INFECTION (Infections and infestations) | 1 (1) | 0 (0)
KLEBSIELLA SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION BACTERIAL (Infections and infestations) | 1 (1) | 0 (0)
ROAD TRAFFIC ACCIDENT (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
STERNAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
LACTIC ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
ARTERIAL THROMBOSIS (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel+Placebo (N=233) | Paclitaxel+ Bevacizumab (N=238)
Anaemia (Blood and lymphatic system disorders) | 39 (82) | 39 (63)
Leukopenia (Blood and lymphatic system disorders) | 14 (42) | 17 (41)
Neutropenia (Blood and lymphatic system disorders) | 50 (124) | 77 (254)
Abdominal pain (Gastrointestinal disorders) | 17 (30) | 20 (27)
Abdominal pain upper (Gastrointestinal disorders) | 13 (14) | 13 (16)
Constipation (Gastrointestinal disorders) | 50 (70) | 67 (108)
Diarrhoea (Gastrointestinal disorders) | 72 (128) | 88 (189)
Dyspepsia (Gastrointestinal disorders) | 16 (20) | 23 (40)
Nausea (Gastrointestinal disorders) | 75 (205) | 99 (310)
Stomatitis (Gastrointestinal disorders) | 26 (35) | 42 (75)
Toothache (Gastrointestinal disorders) | 8 (9) | 15 (16)
Vomiting (Gastrointestinal disorders) | 36 (63) | 47 (96)
Asthenia (General disorders) | 36 (50) | 32 (62)
Fatigue (General disorders) | 74 (123) | 88 (156)
Oedema peripheral (General disorders) | 42 (57) | 41 (56)
Pyrexia (General disorders) | 28 (37) | 34 (59)
Bronchitis (Infections and infestations) | 12 (12) | 11 (14)
Nasopharyngitis (Infections and infestations) | 36 (65) | 24 (54)
Paronychia (Infections and infestations) | 7 (9) | 13 (13)
Upper respiratory tract infection (Infections and infestations) | 11 (14) | 25 (26)
Urinary tract infection (Infections and infestations) | 16 (22) | 35 (47)
Alanine aminotransferase increased (Investigations) | 17 (21) | 21 (37)
Aspartate aminotransferase increased (Investigations) | 16 (19) | 21 (32)
Neutrophil count decreased (Investigations) | 20 (100) | 15 (56)
White blood cell count decreased (Investigations) | 16 (84) | 21 (87)
Decreased appetite (Metabolism and nutrition disorders) | 42 (65) | 55 (91)
Hypokalaemia (Metabolism and nutrition disorders) | 10 (13) | 15 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 53 (86) | 53 (91)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (42) | 26 (32)
Bone pain (Musculoskeletal and connective tissue disorders) | 20 (32) | 11 (17)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (60) | 43 (83)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 (23) | 23 (32)
Dizziness (Nervous system disorders) | 24 (25) | 28 (33)
Dysgeusia (Nervous system disorders) | 22 (24) | 33 (43)
Headache (Nervous system disorders) | 44 (71) | 51 (85)
Neuropathy peripheral (Nervous system disorders) | 50 (67) | 47 (72)
Paraesthesia (Nervous system disorders) | 17 (21) | 12 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 84 (107) | 92 (129)
Anxiety (Psychiatric disorders) | 15 (15) | 8 (8)
Insomnia (Psychiatric disorders) | 20 (24) | 35 (46)
Proteinuria (Renal and urinary disorders) | 26 (33) | 32 (53)
Cough (Respiratory, thoracic and mediastinal disorders) | 30 (38) | 43 (59)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 19 (24)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 (33) | 33 (41)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 48 (77) | 97 (158)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 (15) | 18 (23)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 20 (26)
Alopecia (Skin and subcutaneous tissue disorders) | 145 (159) | 140 (149)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7) | 18 (20)
Nail discolouration (Skin and subcutaneous tissue disorders) | 18 (18) | 33 (37)
Nail disorder (Skin and subcutaneous tissue disorders) | 13 (13) | 13 (14)
Onychomadesis (Skin and subcutaneous tissue disorders) | 6 (6) | 15 (17)
Pruritis (Skin and subcutaneous tissue disorders) | 10 (12) | 15 (17)
Rash (Skin and subcutaneous tissue disorders) | 31 (36) | 58 (113)
Hot flush (Vascular disorders) | 10 (30) | 15 (17)
Hypertension (Vascular disorders) | 30 (83) | 73 (109)
SINUSITIS (Infections and infestations) | 8 (12) | 12 (15)
WEIGHT DECREASED (Investigations) | 5 (5) | 12 (13)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 3 (5) | 12 (13)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 (8) | 12 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.